CLINICAL TRIAL: NCT05744453
Title: The Effect of 12-week Supplementation With Olive Leaf Extract (OLE) on Body Composition and Muscle Strength, Skin-aging and Menopause-related Quality of Life in Postmenopausal Women (45-70 y); a Randomized Controlled Trial
Brief Title: The Effect of 12-week Supplementation With Olive Leaf Extract in Postmenopausal Women (FEMMED)
Acronym: FEMMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioActor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NL81363.068.22
Record Dates: First submitted 2022-12-08; First posted 2023-02-27 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Post-Menopausal Women
Keywords: Post-Menopause; Body composition; Supplementation
MeSH Terms: interventions — olive leaf extract; Cellulose

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Block Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive Leaf Extract (Experimental): Olive leaf extract supplementation
  Interventions: Dietary Supplement: Olive Leaf Extract
- Control (Placebo Comparator): Cellulose Supplementation
  Interventions: Dietary Supplement: Cellulose

INTERVENTIONS:
Dietary Supplement: Olive Leaf Extract — experimental arm
  Arms: Olive Leaf Extract
Dietary Supplement: Cellulose — placebo comparator arm
  Arms: Control

SUMMARY:
Menopause is defined as the end of menstruation and fertility,starting 12 months after the last menstrual period.In this modern and economically developed society, most women are living for at least 20-40 years in a postmenopausal state. During menopause women may experience physical, emotional, and urogenital symptoms, with a significant impact on their health.Olive leaf extract supplementation may improve quality of life in post-menopausal women.

DETAILED DESCRIPTION:
Menopause is associated with abdominal adipose tissue accumulation and the loss of muscle mass which causes a decrease in muscle strength. Moreover, the decrease in estrogens associated with menopause increases the risk of osteoporosis. The supplementation of oleuropein, the most abundant polyphenol found in olive tree leaves, can be an effective strategy to ameliorate body composition, due to its potential to attenuate the aging-induced decrease in protein content in muscles, to enhance thermogenesis in adipose tissue and to increase serum osteocalcin, a bone turnover marker. The current study wants to investigate the effect of 12-week olive leaf extract supplementation on body composition and muscle strength, skin-aging and menopause-related quality of life in postmenopausal women (45-70 y).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (amenorrhea over 12 months)
* Age between 45-70 years
* Body mass index (BMI) < 35 kg/m2

Exclusion Criteria:

* Use of hormone replacement therapy (estrogenic or progestogenic) in the past 3 months before T1
* Allergy to test product/control or olive leaves/olive oil
* Use of antibiotics within 3 months prior T1
* Use of probiotics or supplements containing vitamins,minerals or antioxidants four weeks prior T1 (Calcium and vitamin D supplementation are permitted)
* Use of isoflavone-derived supplements four weeks prior T1
* Regular smoking (including use of e-cigarettes)
* Abuse of alcohol (alcohol consumption >20 units/week) and/or drugs
* Intention to take part in any weight loss program
* Underwent Botulinum toxin A (Botox) injection treatment near the test sites within 2 years of baseline or plan to receive this treatment during the study
* Underwent Filler injection (collagen, hyaluronic acid, etc.) near the test sites within 2 years of baseline or plan to receive this treatment during the study
* Not willing to avoid over exposure to sun or tanning session (solarium) on the test area within 30 days prior to study start and for the duration of the study (exposure after application of sunscreen allowed)
* Willing not to change the routine use of facial cream/treatment during the study duration
* Treatment with an investigational drug (phase 1-3) 180 days before the start of the study
* Diagnosed with medical conditions that might interfere with endpoints or compromise participant safety during testing (e.g. Cardiovascular diseases, diabetes, skin diseases, cancer, Parkinson's disease, Gastrointestinal diseases or abdominal surgery interfering with gastrointestinal function) to be decided by the principal investigator
* Medication intake that might interfere with endpoints or compromise participant safety during testing (e.g. Glucose-Lowering Medications such as Metformin) to be decided by the principal investigator

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-Menopausal Symptoms
Enrollment: 65 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Changes in body composition (total and regional fat mass and fat free mass) measured using Dual-energy X-ray absorptiometry (DXA) | At baseline + after 12 weeks of supplementation
  Quantified through Dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Evaluate changes in muscle strength between study product and placebo groups | At baseline + after 6 weeks + after 12 weeks of supplementation
  Measured by a calibrated hand dynamometer.
Evaluate changes in skin health between study product and placebo groups | At baseline + after 6 weeks + after 12 weeks of supplementation
  Measured by a visual analogue scale (VAS)
Evaluate changes in menopause-related symptoms between study product and placebo groups | At baseline + after 6 weeks + after 12 weeks of supplementation
  Measured by a quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Troost, Dr, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lasfar A, van Stratum SLM, Imperatrice M, van Kalkeren CAJ, Scheijen JLJM, Schalkwijk CG, La Torre D, Troost FJ. Effects of olive leaf extract supplementation on systemic markers of tissue aging and remodeling in postmenopausal women: a randomized controlled trial with exploratory skin outcomes. Front Nutr. 2025 Nov 18;12:1670194. doi: 10.3389/fnut.2025.1670194. eCollection 2025. PMID 41340653